CLINICAL TRIAL: NCT05074667
Title: Use of Continuous Glucose Monitors in Publicly-Insured Youth With Type 2 Diabetes - A Pilot and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sejal Shah, Clinical Assistant Professor of Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 62166
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous Glucose Monitor (Other): All participants will be included in this arm
  Interventions: Device: Continuous Glucose Monitor; Other: Patient Reported Outcome Questionnaires

INTERVENTIONS:
Device: Continuous Glucose Monitor — Participants will be provided a continuous glucose monitor for use in self-glucose monitoring as per standard clinical care
Other: Patient Reported Outcome Questionnaires — Participants and their parents will be asked to complete patient reported outcome questionnaires at 3 study time points.

SUMMARY:
The purpose of this pilot feasibility study is to provide continued CGM access to youth with type 2 diabetes and collect descriptive data about feasibility of use of CGM in youth with type 2 diabetes ages 4 years and older. From this study the investigators hope to learn if CGM use in youth with type 2 diabetes can be tolerated and sustained with good adherence and to describe blood glucose patterns in youth with type 2 diabetes. The primary aim will be to evaluate the feasibility of CGM start and continuation in youth with T2D and describe glucose metrics and patient reported outcomes (PROs). The investigators will pilot and refine a program to test the hypothesis that CGM start and continuation in youth with T2D is feasible and then evaluate glucose metrics and PROs.

ELIGIBILITY:
Inclusion Criteria:

* public insurance
* between ages 4-19.99 years inclusive
* diagnosis of T2D (diabetes autoantibody negative) followed in the Pediatric Endocrinology clinic at Stanford Children's Health
* HbA1C greater than 6.5% at enrollment
* interested in starting on a continuous glucose monitor
* have access to a mobile device that is compatible with CGM applications or willing to use CGM receiver provided

Exclusion Criteria:

* non-T2D diagnosis
* HgA1C < 6.5%
* are not willing to wear CGM
* have private health insurance.

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sejal Shah, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Children's Health, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal, for purpose of achieving aims in the approved proposal. Proposals should be directed to the protocol director and data sharing requests will need to follow current protocols in place at Stanford University.

REFERENCES:
- [Derived] Shah S, Tanenbaum ML, Loyola A, Sala NGL, Darji H, Hanes S, Bishop FK, Hood KK, Maahs DM. Use of Continuous Glucose Monitors in Publicly Insured Youth With Type 2 Diabetes: A 12-month Pilot and Feasibility Study. J Diabetes Sci Technol. 2025 Sep 20:19322968251368366. doi: 10.1177/19322968251368366. Online ahead of print. PMID 40974209
- See also: PROMIS scoring manual — https://www.healthmeasures.net/images/PROMIS/manuals/Scoring_Manuals_/PROMIS_Global_Health_Scoring_Manual.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Glucose Monitor: Participants are provided a continuous glucose monitor for use in self-glucose monitoring as per standard clinical care. Participants and their parents are asked to complete patient reported outcome questionnaires at 3 study time points.
Period: Overall Study
Arm/Group | Continuous Glucose Monitor
Started | 30
Completed | 15
Not Completed | 15
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.19 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian and Pacific Islander | 1
  Hispanic | 27
  Non Hispanic Black | 1
  Non Hispanic White | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 75% Wear Time Over 14 Days as a Measure of Sustained CGM Use
Time Frame: months 2,3,6,9 and 12 (assessed over the 14 days prior to each clinic visit)
Population: Participants with available CGM data at each respective timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 24
Participants
  2-month visit | 7
  3-month visit: number analyzed (Participants) | 15
  3-month visit | 2
  6-month visit: number analyzed (Participants) | 14
  6-month visit | 1
  9-month visit: number analyzed (Participants) | 10
  9-month visit | 0
  12-month visit: number analyzed (Participants) | 7
  12-month visit | 0

2. Secondary Outcome: Mean HbA1C
Description: HbA1C through 12 months of CGM use
Time Frame: baseline and months 2,3,6,9 and 12
Population: Participants with available data at each respective timepoint
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 30
percentage of glycosylated hemoglobin
  baseline | 10.18 (2.65)
  2-month visit: number analyzed (Participants) | 24
  2-month visit | 10.16 (2.69)
  3-month visit: number analyzed (Participants) | 15
  3-month visit | 8.95 (2.91)
  6-month visit: number analyzed (Participants) | 14
  6-month visit | 9.27 (2.71)
  9-month visit: number analyzed (Participants) | 10
  9-month visit | 10.04 (2.214)
  12-month visit: number analyzed (Participants) | 7
  12-month visit | 9.77 (1.22)

3. Secondary Outcome: Time With Glucose Values in Target Range of 70-180 mg/dL
Time Frame: months 2,3,6,9 and 12 (assessed over the 14 days prior to each clinic visit)
Population: Participants with available CGM data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 24
percentage of time
  2-month visit | 71 [18 to 93.25]
  3-month visit: number analyzed (Participants) | 15
  3-month visit | 45.5 [11.25 to 87.75]
  6-month visit: number analyzed (Participants) | 14
  6-month visit | 59 [37 to 86]
  9-month visit: number analyzed (Participants) | 10
  9-month visit | 28.5 [7.5 to 53.75]
  12-month visit: number analyzed (Participants) | 7
  12-month visit | 42 [31 to 77]

4. Secondary Outcome: PROMIS Global Health Overall Scale Score
Description: PROMIS Global Health (7 questions, Minimum=1, maximum=5 for each question, higher score for physical health questions is better outcome, higher score for mental health is worse outcome). Scores for each question were summed then converted to a t-score (overall range 16 to 67.5, higher score = better health). A score of 50 is the average for the United States general population with a standard deviation of 10. A score below 22 in this study would result in a referral to social work or diabetes psychology.
Time Frame: baseline, months 3 and 12
Population: Participants with available data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 30
T-score
  baseline | 37.20 [30.00 to 40.40]
  3-month visit: number analyzed (Participants) | 14
  3-month visit | 35.60 [32.40 to 38.80]
  12-month visit: number analyzed (Participants) | 12
  12-month visit | 32.40 [29.20 to 35.60]

5. Secondary Outcome: PedsQL 3.2 Overall Scale Score - Participant Rated
Description: Pediatric Quality of Life Inventory (PedsQL) Diabetes Module version 3.2, including 33 items (questions) comprising 5 dimensions (diabetes symptoms, treatment 1, treatment 2, worry, and communication). Each item scored from 0 to 4, higher scores correspond to lower problems. Each item is reversed scored and linearly transformed to a 0 to 100 scale (0=100,1=75,2=50,3=25,4=0), higher scores correspond to lower problems. The overall score is calculated as the sum of the transformed scores for each item divided by the total number of items answered by participants to create an overall score range of 0 to 100, higher scores correspond to lower problems.
Time Frame: baseline and months 3 and 12
Population: Participants with available data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 30
score on a scale
  Peds QL Diabetes - baseline | 58.33 [50.00 to 71.67]
  Peds QL Diabetes - month 3: number analyzed (Participants) | 14
  Peds QL Diabetes - month 3 | 65.00 [55.83 to 72.92]
  Peds QL Diabetes - month 12: number analyzed (Participants) | 12
  Peds QL Diabetes - month 12 | 58.33 [45.00 to 69.58]
  Peds QL Overall - baseline | 65.53 [58.33 to 71.97]
  Peds QL Overall - month 3: number analyzed (Participants) | 14
  Peds QL Overall - month 3 | 59.85 [56.82 to 72.92]
  Peds QL Overall - month 12: number analyzed (Participants) | 12
  Peds QL Overall - month 12 | 55.30 [52.84 to 65.72]

6. Secondary Outcome: PedsQL 3.2 Scale Score - Parent Rated
Description: Pediatric Quality of Life Inventory (PedsQL) Diabetes Module version 3.2, including 33 items (questions) comprising 5 dimensions (diabetes symptoms, treatment 1, treatment 2, worry, and communication). Each item scored from 0 to 4, higher scores correspond to lower problems. Each item is reversed scored and linearly transformed to a 0 to 100 scale (0=100,1=75,2=50,3=25,4=0), higher scores correspond to lower problems. The overall score is calculated as the sum of the transformed scores for each item divided by the total number of items answered by parents to create an overall score range of 0 to 100, higher scores correspond to lower problems. Parents completed the survey at the same time as their child but were not considered to be enrolled in the study.
Time Frame: baseline and months 3 and 12
Population: Participants with available data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 19
score on a scale
  Peds QL Diabetes - baseline | 65.00 [61.67 to 73.33]
  Peds QL Diabetes - month 3: number analyzed (Participants) | 11
  Peds QL Diabetes - month 3 | 60.00 [55.83 to 68.33]
  Peds QL Diabetes - month 12: number analyzed (Participants) | 14
  Peds QL Diabetes - month 12 | 59.17 [54.58 to 72.08]
  Peds QL Overall - baseline | 64.39 [56.06 to 70.76]
  Peds QL Overall - month 3: number analyzed (Participants) | 11
  Peds QL Overall - month 3 | 59.85 [50.76 to 68.94]
  Peds QL Overall - month 12: number analyzed (Participants) | 14
  Peds QL Overall - month 12 | 57.58 [52.84 to 73.86]

7. Secondary Outcome: Diabetes Technology Attitudes (DTA) - Participant Rated
Description: The DTA assesses use and comfort with technology. Each of the 5 items are responded to on a 5 point likert scale (from 1=Strongly Disagree to 5=Strongly Agree) Mean item score, higher score = more positive attitude, total score range 1-5
Time Frame: 1 year (assessed at baseline, 3 months and 12 months)
Population: Participants with available data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 28
score on a scale
  baseline | 3.78 [3.55 to 4.25]
  3-month visit: number analyzed (Participants) | 14
  3-month visit | 4.50 [3.65 to 4.95]
  12-month visit: number analyzed (Participants) | 12
  12-month visit | 4.00 [3.75 to 4.55]

8. Secondary Outcome: Diabetes Technology Attitudes (DTA) - Parent Rated
Description: The DTA assesses use and comfort with technology. Each of the 5 items are responded to on a 5 point likert scale (from 1=Strongly Disagree to 5=Strongly Agree) Mean item score, higher score = more positive attitude, total score range 1-5 Parents completed the survey at the same time as their child but were not considered to be enrolled in the study.
Time Frame: 1 year (assessed at baseline, 3 months and 12 months)
Population: Participants with available data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 19
score on a scale
  baseline | 3.80 [3.40 to 3.80]
  3-month visit: number analyzed (Participants) | 11
  3-month visit | 4.00 [3.60 to 4.50]
  12-month visit: number analyzed (Participants) | 16
  12-month visit | 3.60 [3.35 to 4.05]

9. Secondary Outcome: Problem Areas in Diabetes-Teen Version (PAID-T) Overall Scale Score - Participant Rated
Description: Problem Areas in Diabetes - survey Teen version with 14 questions each scored using a 6-point Likert Scale (1=not a problem, to 6=serious problem). The overall score is computed by summing responses for an overall range of 14 to 84 (higher score is worse outcome).
Time Frame: baseline, months 3 and 12
Population: Participants who completed the PAID Teen survey
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 20
score on a scale
  baseline | 43.50 [30.75 to 47.00]
  3-month visit | 47.00 [34.25 to 62.50]
  12-month visit | 52.00 [40.50 to 60.50]

10. Secondary Outcome: Problem Areas in Diabetes (P-PAID) Overall Scale Score - Parent Rated
Description: Problem Areas in Diabetes - survey Teen Parent version with 15 questions each scored using a 6-point Likert Scale (1=not a problem, to 6=serious problem). The overall score is computed by summing responses for an overall range of 15 to 90 (higher score is worse outcome). Parents completed the survey at the same time as their child but were not considered to be enrolled in the study.
Time Frame: baseline, months 3 and 12
Population: Participants with available data at each respective timepoint
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitor
Number analyzed (Participants) | 19
score on a scale
  baseline | 55.00 [46.00 to 69.50]
  3-month visit: number analyzed (Participants) | 11
  3-month visit | 59.00 [48.50 to 69.00]
  12-month visit: number analyzed (Participants) | 14
  12-month visit | 50.50 [42.75 to 68.00]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Continuous Glucose Monitor
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05074667/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT05074667/ICF_000.pdf